CLINICAL TRIAL: NCT04142450
Title: CoolSculpting® the Upper Arms and Inner Thighs in Participants of Chinese Descent (XinCOOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-MA-PLS-0633
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Masking Description: This is an open-label study. Blinding will only be employed for photograph review by an independent panel of physician reviewers with expertise in the areas of dermatology and/or plastic surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CoolSculpting® System (Experimental): Participants underwent a single CoolSculpting® treatment session on Day 1 that was comprised of timed segments of cooling followed by 2 minutes of manual massage. Each treated arm had up to two timed segments (or cycles) in the treatment session, each treated thigh had one timed segment (or cycle) in the treatment session.
  Interventions: Device: CoolSculpting® System

INTERVENTIONS:
Device: CoolSculpting® System — Each participant underwent a single treatment session that was comprised of timed segments of cooling followed by 2 minutes of manual massage.

SUMMARY:
To evaluate the safety and effectiveness of the Allergan CoolSculpting® system using CoolAdvantage applicators for non-invasive subcutaneous fat reduction of the upper arms and inner thighs in participants of Chinese descent.

ELIGIBILITY:
Inclusion Criteria:

* Participant (healthy volunteers) has read and signed the study written informed consent form (ICF)
* 1st or 2nd generation, non-mixed race, Chinese descent.
* Participant has clearly visible and palpable fat on the left and right lower aspects of the upper arms and/or left and right inner thighs, which in the investigator's opinion is appropriate and may benefit from the treatment.
* Participant has not had weight change fluctuations exceeding 4.5 kilograms (kg) (or 5% of body weight) in the preceding month.
* Participant has a body mass index (BMI) of ≥ 18.5 to ≤ 30. A BMI is defined as weight in kilograms divided by height in meters squared (kg/m^2).
* Participant agrees to maintain weight (i.e., within 5% of body weight) by not making any changes in diet or exercise routine during the course of the study.
* Participant agrees to have photographs taken of the treatment area(s) during the scheduled time periods.

Exclusion Criteria:

* Participant has a history of an invasive fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.), or implants in or immediately adjacent to the area of intended treatment.
* Participant has a history of prior surgery or scar tissue on the arms and/or inner thighs related to the area being considered for treatment.
* Participant has a known history of cryoglobulinemia, cold urticaria, cold agglutinin disease, or paroxysmal cold hemoglobinuria.
* Participant has a known sensitivity to cold or has any condition with a known response to cold exposure that limits blood flow to the skin, such as cold urticaria, Raynaud's disease, or Chilblains (pernio).
* Participant with a clinically significant bleeding disorder, or concomitant use of oral or subcutaneous anticoagulants, or is taking any medication that in the investigator's opinion may significantly increase the participant's risk of bruising.
* Participant with a history of carpal tunnel syndrome, compartment syndrome, or deep vein thrombosis in the upper or lower extremities.
* Participant is currently taking or has taken diet pills or weight control supplements within the past 6 months.
* Participant has any dermatological conditions, such as moderate to excessive skin laxity, infection, open wound, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks are not an exclusion).
* Participant has an active implanted device such as a pacemaker, defibrillator, drug delivery system, or any other metal-containing implant within or adjacent to the area being considered for treatment.
* Participant is pregnant or intending to become pregnant in the next 3 months.
* Participant is lactating or has been lactating in the past 6 months.
* Participant is unable or unwilling to comply with the study requirements.
* Participant is currently enrolled in a clinical study of any unapproved investigational device, investigational product, or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participant has any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the participant's response or the integrity of the data or would pose an unacceptable risk to the participant.
* Participant has had a non-invasive fat reduction and/or body contouring procedure in the area(s) of intended treatment within the past 12 months.
* Participant needs to administer, or has a known history of subcutaneous injections, into the area(s) of intended treatment (e.g., cortisone, heparin, insulin) within the past 6 months.
* Participant with known sensitivity or allergy to fructose, glycerin, isopropyl alcohol, or propylene glycol.
* Participant with impaired peripheral circulation in the area to be treated.
* Participant with neuropathic disorders such as post-herpetic neuralgia or diabetic neuropathy.
* Participant with impaired skin sensation.
* Participant with a history of hernia in or adjacent to the treatment area(s) site.
* Participant with a skin condition such as eczema, dermatitis, or rashes in the area to be treated.
* Participant diagnosed with a systemic fibrosing disease or fibrosis in the area intended or adjacent to the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hickling, Study Director — Allergan
Locations (3):
- Canada (3):
  - Vancouver Laser and Skin Care Clinic, Vancouver, British Columbia
  - Project Skin MD, Vancouver, British Columbia
  - Pacific Derm, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. — http://www.AllerganClinicalTrials.com
- See also: To be considered as a site for current and future Allergan Clinical Trials, please register using the Investigator Databank link. — http://www.investigatordatabank.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CoolSculpting® System
Started | 50
Safety Population (Safety Population included all treated participants.) | 49
Completed | 48
Not Completed | 2
Not completed — Screen Failure | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all treated participants.
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  First Generation, Non-Mixed Chinese | 22
  Second Generation, Non-Mixed Chinese | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Arms With Correct Identification of Baseline Versus 12-week Treatment Images of the Upper Arms by at Least Two Out of Three Blinded, Independent Reviewers
Description: Baseline versus 12-week images of the participants' left and right upper arms were assessed separately by the reviewers. Success was defined as at least 75% correct identification of the pre-treatment images of the upper arms.
Time Frame: Baseline (Day 1) to Week 12
Population: Per Protocol Population, consisted of all treated participants followed for 12 weeks and with weight change of no more than 5% of total body weight at the time the 12-week images were taken. Overall number analyzed are the number of participants and number of arms treated per protocol with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of arms
Units Other Than Participants: arms
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 36
Number analyzed (arms) | 72
percentage of arms | 76.4 [64.9 to 85.6]

2. Secondary Outcome: Percentage of Thighs With Correct Identification of Baseline Versus 12-week Treatment Images of the Inner Thighs by at Least Two Out of Three Blinded, Independent Reviewers
Description: Baseline versus 12-week images of the participants' left and right thighs were assessed separately by the reviewers. Success was defined as at least 75% correct identification of the pre-treatment images of the inner thighs.
Time Frame: Baseline (Day 1) to Week 12
Population: Per Protocol Population consisted of all treated participants followed for 12 weeks and with weight change of no more than 5% of total body weight at the time the 12-week images were taken. Overall number analyzed are the number of participants and number of thighs treated per protocol with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of thighs
Units Other Than Participants: thighs
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 20
Number analyzed (thighs) | 40
percentage of thighs | 70.0 [53.5 to 83.4]

3. Secondary Outcome: Number of Participants With a Response of 'Satisfied' or 'Very Satisfied' for Question 1 (Overall Satisfaction) on the CoolSculpting Participant Questionnaire at the 12-week Visit for the Upper Arms
Description: Participants were asked to complete a survey upon completing the treatment to assess their level of satisfaction with the treatment. Participants selected one of five options: 'very satisfied', 'satisfied', 'neither satisfied nor dissatisfied', 'dissatisfied', or 'very dissatisfied'.
Time Frame: Week 12
Population: Per Protocol Population consisted of all treated participants followed for 12 weeks and with weight change of no more than 5% of total body weight at the time the 12-week images were taken. Number of participants analyzed are the number of participants with arms treated with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 36
Participants | 22

4. Secondary Outcome: Number of Participants With a Response of 'Satisfied' or 'Very Satisfied' for Question 1 (Overall Satisfaction) on the CoolSculpting Participant Questionnaire at the 12-week Visit for the Inner Thighs
Description: as for outcome 3
Time Frame: Week 12
Population: Per Protocol Population consisted of all treated participants followed for 12 weeks and with weight change of no more than 5% of total body weight at the time the 12-week images were taken. Number of participants analyzed is the number of participants with thighs treated with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 40
Participants | 26

5. Secondary Outcome: Change From Baseline in Mean Fat Reduction Using Caliper Measurements at Week 12 for Upper Arms
Description: Caliper measurements of the treatment areas were taken at baseline and at 12-weeks post treatment. After the treatment area was identified and marked, the thickness of the fat layer was measured using a caliper at the middle of the fat bulge. For each treatment area, three measurements were taken and recorded. The average of the three measurements was calculated. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: Per Protocol Population consisted of all treated participants followed for 12 weeks and with weight change of no more than 5% of total body weight at the time the 12-week images were taken. Overall number analyzed are the number of participants and number of arms treated per protocol with data available for analyses.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Units Other Than Participants: arms
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 36
Number analyzed (arms) | 72
millimeter (mm)
  Baseline (Day 1) | 26.7 (5.54)
  Change from Baseline to Week 12 | -7.0 (5.72)

6. Secondary Outcome: Change From Baseline in Mean Fat Reduction Using Caliper Measurements at Week 12 for Inner Thighs
Description: as for outcome 5
Time Frame: Baseline (Day 1) to Week 12
Population: Per Protocol Population consisted of all treated participants followed for 12 weeks and with weight change of no more than 5% of total body weight at the time the 12-week images were taken. Overall number analyzed are the number of participants and number of thighs treated per protocol available for analyses.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: thighs
Arm/Group | CoolSculpting® System
Number analyzed (Participants) | 40
Number analyzed (thighs) | 80
mm
  Baseline (Day 1) | 32.2 (9.28)
  Change from Baseline to Week 12 | -4.3 (12.44)

ADVERSE EVENTS:
Time Frame: Day 1 Treatment to Week 12 +/- 14 days
Description: Protocol provided an extensive, detailed list of well-known anticipated device effects which were not considered adverse events (AEs) unless severity caused disruption to the participant's daily activities, or lasted longer than anticipated duration, in which case they were evaluated as potential AEs. Safety Population included all treated participants.
Arm/Group | CoolSculpting® System
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04142450/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04142450/SAP_001.pdf